CLINICAL TRIAL: NCT05105165
Title: Correlation Between Serum Orphanin FQ and β1-AR Autoantibodies in Patients With Chronic Ischemic Heart Failure and Its Regulatory Mechanism
Brief Title: Regulatory Mechanism of Orphanin FQ in Patients With Chronic Ischemic Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, Director, Second Hospital of Shanxi Medical University
Other Study IDs: hanyi20210623
Record Dates: First submitted 2021-07-04; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Antibody positive group
  Interventions: Diagnostic Test: Enzyme linked immunosorbent assay
- Antibody negative group
  Interventions: Diagnostic Test: Enzyme linked immunosorbent assay
- Health Group
  Interventions: Diagnostic Test: Enzyme linked immunosorbent assay

INTERVENTIONS:
Diagnostic Test: Enzyme linked immunosorbent assay — Determination of serum β 1-aa content

SUMMARY:
β 1 adrenergic autoantibody on cardiomyocytes β 1 adrenergic receptor increased the occurrence of malignant arrhythmia in patients with chronic heart failure, accelerated myocardial cell damage, and participated in sudden cardiac death. Our team found for the first time that endogenous orphanin enkephalin promotes arrhythmia after acute myocardial ischemia in rats, and its mechanism includes PKC pathway, regulation of action potential duration and cell membrane surface β 1 adrenoceptor internalization disorder. At the same time, N / OFQ can regulate the level of immune factors, and immune factors participate in the formation of β1-aa. This study will be verified by clinical observation and animal experiments: first, N / OFQ, IL-6 and chronic ischemic heart failure, and β 1-aa; second, relationship between IL-6 gene 572G / C polymorphism and chronic ischemic heart failure correlation of β 1-aa production; last, objective to verify whether N / OFQ is involved in the regulation of IL-6 on chronic ischemic heart failure by knocking out N/ OFQ gene in the animal model of chronic ischemic heart failure. So as to clarify the mechanism of myocardial cell and extracellular injury, and find a new target for the treatment of chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure patients with reduced ejection fraction due to ischemic heart disease.

Exclusion Criteria:

* Restrictive or hypertrophic cardiomyopathy, hypertensive cardiomyopathy, acute myocarditis, acute coronary syndrome or acute myocardial infarction in the last 2 months, valvular disease (except mitral regurgitation secondary to left ventricular dilation).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: During the study period, patients in the Department of Cardiology of the second hospital of Shanxi Medical University were admitted.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11-28 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum orphanin FQ was determined by enzyme linked immunosorbent assay | 24 hours
  Serum N/OFQ levels

IPD SHARING:
Plan to Share IPD: No